CLINICAL TRIAL: NCT04475887
Title: Treatment of Anemia With Intravenous Iron in Patients Listed for Orthotopic Liver Transplantation
Acronym: TRAILER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Georg Gyoeri, Head of Liver Transplantation Outpatient Clinic, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1175/2017
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Liver Transplantation; Blood Loss
Keywords: liver; anemia; transplantation
MeSH Terms: conditions — Hemorrhage; Anemia | interventions — ferric carboxymaltose; Iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): IV administration of iron-III-carboxymaltose according to iron deficit every 4 weeks.
  Interventions: Drug: Iron Carboxymaltose
- Group B (Placebo Comparator): IV administration of 1000ml 0.9% NaCl every 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iron Carboxymaltose — see above
  Other Names: IRON
  Arms: Group A
Drug: Placebo — see above
  Arms: Group B

SUMMARY:
The aim of this study is to investigate whether therapy with intravenous iron carboxymaltose in patients with iron deficiency anemia (IDA) listed for orthotopic liver transplantation (OLT) increases hemoglobin concentrations and reduces intraoperative transfusion of packed red blood cells (PRBCs). The investigators hypothesize that therapy with intravenous iron will increase hemoglobin concentrations and reduce intraoperative transfusion of PRBCs in patients with IDA listed for OLT.

ELIGIBILITY:
Inclusion Criteria:

* patients listed for OLT with positive screening for IDA

Exclusion Criteria:

* Age <18 years
* Hemochromatosis
* Iron utilization disorders
* Non-IDA
* Therapy with erythropoietin-stimulating agents or intravenous iron within 4 weeks prior to screening
* Previous allergic reactions against intravenous iron formulations
* Transfusion within 2 weeks prior to screening
* Complete portal vein thrombosis
* High-urgency OLT
* Pregnancy
* Sepsis or severe infection
* Immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-23 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin at OLT | 6 months
  Change in hemoglobin concentrations from baseline until before induction of anesthesia for OLT

SECONDARY OUTCOMES:
Transfusion requirement | 6 months
  Transfusion of PRBCs during and within the first 24 hours following OLT
Hemoglobin after 4 weeks | 4 weeks
  Change in hemoglobin concentrations from baseline until 4 weeks after initiation of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Georg P Gyoeri, MD, Principal Investigator — Department of Surgery; David M Baron, MD, Principal Investigator — Department of Anaesthesiology
Locations (1):
- Medical University of Vienna, Department of Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No